CLINICAL TRIAL: NCT01328236
Title: Bortezomib in Combination With Liposomal Doxorubicin and Dexamethasone to Treat Plasma Cell Leukemia
Acronym: Bortezomib
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Service, China (Industry)
Collaborators: Harbin Hematology and Oncology Institute (Other); Shanghai Changzheng Hospital (Other); Chinese PLA General Hospital (Other); 307 Hospital of PLA (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Beijing Chao Yang Hospital (Other); Henan Provincial People's Hospital (Other); Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, wangzhao, Beijing Friendship Hospital, Clinical Service, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26866138CAN2026; NCT01327716 (obsolete NCT alias)
Record Dates: First submitted 2011-03-29; First posted 2011-04-04 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Plasma Cell Leukemia; Multiple Myeloma
Keywords: Bortezomib; PCL
MeSH Terms: conditions — Leukemia, Plasma Cell; Multiple Myeloma | interventions — Bortezomib; liposomal doxorubicin; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- V-DD single arm (Experimental): INDUCTION THERAPY: V-DD induction therapy for 6 cycles，28 Days per Cycle. Bortezomib - 1.3 mg/m2 IV, Days 1, 4, 8 , 11 of every treatment; Liposomal Doxorubicin - 30 mg/m2 IV, Day 4 of every treatment; Dexamethasone - 40 mg/d IV, Days 1 - 4 of every treatment.
  Maintenance treatment for 4 cycles,28 Days per Cycle. Thalidomide - 100mg Qn ; Bortezomib - 1.3 mg/m2 IV ,Days 1, 4, 8 and 11 of every treatment; Dexamethasone - 40 mg/d IV ,Days 1 - 4; Interferon - 300 u Qod,（Specially for IgA type）. Interval between every two cycles for 6 months, until progression or unacceptable toxicity develops.
  Interventions: Drug: Bortezomib; Drug: Liposome doxorubicin; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bortezomib — INDUCTION THERAPY: 1.3 mg/m2, IV (in the vein) on day 1， 4， 8， 11 of each 28 day cycle. 6 Cycles: until progression or unacceptable toxicity develops.
  MAINTENANCE THERAPY: 1.3 mg/m2, IV (in the vein) on day 1， 4， 8， 11 of each 28 day cycle. 4 Cycles: interval between every two cycles for 6 months, until progression or unacceptable toxicity develops.
  Other Names: Velcade
Drug: Liposome doxorubicin — INDUCTION THERAPY: 30 mg/m2, IV (in the vein) on day 4 of each 28 day cycle. 6 Cycles: until progression or unacceptable toxicity develops.
  Other Names: Caelyx
Drug: Dexamethasone — INDUCTION THERAPY: 40 mg/d, IV (in the vein) on day 1- 4 of each 28 day cycle. 6 Cycles: until progression or unacceptable toxicity develops.
  MAINTENANCE THERAPY: 40 mg/d, IV (in the vein) on day 1- 4 of each 28 day cycle. 4 Cycles: interval between every two cycles for 6 months, until progression or unacceptable toxicity develops.
  Other Names: Acidocont, Deronil, Dexacortal, dexametona, Flumeprednisolon

SUMMARY:
Bortezomib/Liposomal doxorubicin (V-DD) is preferred to bortezomib single agent in salvage therapy for Multiple Myeloma (MM).

The present study is designed to assessment the efficacy and safety study of Bortezomib in combination with Liposomal Doxorubicin and Dexamethasone in treatment of Plasma Cell Leukemia (PCL).

Primary study endpoint is the overall response rate (sCR+CR+VGPR+PR). Secondary endpoints is the rate of complete response (sCR+CR), partial remission rate (VGPR + PR), duration of response (DOR), overall survival (OS).

DETAILED DESCRIPTION:
Patient with Plasma Cell Leukemia(PCL ) and multiple myeloma (MM); KPS ≥ 60scores

ELIGIBILITY:
Inclusion Criteria:

* Patients confirmed relapsed or refractory PCL who previously untreated or never received treatment with Bortezomib
* KPS ≥ 60
* Adequate liver and renal function within 2 weeks of Screening:
* Bilirubin ≤ 1.5 × the upper limit of normal (ULN)
* Alanine aminotransferase (ALT) ≤ 2.5 × the upper limit of normal (ULN)
* Aspartate aminotransferase (AST) ≤ 2.5 × the upper limit of normal (ULN)
* Cardiac function > Ⅲ grade and ejection fraction > 45%
* Signed informed consent prior to initiation of any study-related procedures that are not considered standard of care

Exclusion Criteria:

* has taken Bortezomib
* KPS ≤ 60 scores
* mental illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
overall response rate | Day 1 of every treatment cycle
  The overall response rate of V-DD in patients with PCL assessed by International Myeloma Working Group(IMWG) criteria

SECONDARY OUTCOMES:
the rate of response | Day 1 of every treatment cycle
  The complete response rate of V-DD in patients with PCL assessed by International Myeloma Working Group(IMWG) criteria.
partial remission rate | Day 1 of every treatment cycle
  The complete response rate of V-DD in patients with PCL assessed by International Myeloma Working Group(IMWG) criteria.
duration of response | up to 6 months
overall survival | up to two and a half year
Adverse Events | up to two and a half years
  Occurrence of adverse events throughout the study using CTCAE ctriteria version 4.0.
FACT/GOC-Ntx | Day 1 of every treatment cycle

CONTACTS AND LOCATIONS:
Overall Officials: zhao wang, Master, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Clinical Service Center, Beijing, Beijing Municipality, China